CLINICAL TRIAL: NCT06751745
Title: Effectiveness of Online Emotional Intelligence Training Among Bangladeshi Youths: A Quasi-Experimental Study
Brief Title: Effectiveness of Online Emotional Intelligence Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bangladesh Institute of Innovative Health Research (Other)
Responsible Party: Principal Investigator, Faisal Ahmed, Research Coordinator, Bangladesh Institute of Innovative Health Research
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BIIHR-2024-007
Record Dates: First submitted 2024-12-20; First posted 2024-12-30 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-12

CONDITIONS: Emotional Intelligence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental)
  Interventions: Behavioral: Online Emotional Intelligence Training

INTERVENTIONS:
Behavioral: Online Emotional Intelligence Training — The intervention is a 4-week online Emotional Intelligence (EI) training program for Bangladeshi youth. It includes weekly one-hour sessions focusing on self-awareness, self-regulation, social awareness, and relationship management. Led by experts, the program uses interactive activities and practical exercises to enhance emotional skills. Pre- and post-training assessments with the Bengali Emotional Intelligence Scale measure outcomes.

SUMMARY:
The proposed study, titled "Effectiveness of Emotional Intelligence Training among Bangladeshi Youth," aims to evaluate the impact of a 4-week online Emotional Intelligence (EI) training program on the emotional competencies of Bangladeshi youth. Emotional intelligence, which encompasses skills such as self-awareness, self-regulation, social awareness, and relationship management, is crucial for personal and professional success, as well as mental well-being.

The study hypothesizes that targeted EI training can enhance emotional competencies, leading to improved social skills, decision-making, and mental health outcomes. This is particularly significant in the Bangladeshi context, where such programs are scarce, and youth face numerous societal pressures. The research will employ a quantitative, experimental design, comparing pre- and post-training EI levels between an experimental group (participants undergoing EI training) and a control group (participants not receiving the training).

Participants, aged 18 to 30 years, will be recruited from educational institutions across Bangladesh. The study will use the Bengali version of the Emotional Intelligence Scale to assess EI levels and a structured Personal Information Form to collect demographic data. The training program will consist of four weekly sessions, each focusing on a core EI component: self-awareness, self-regulation, social awareness, and relationship management. The sessions will be conducted by experts in public health and psychology.

Data analysis will involve descriptive statistics, t-tests, and regression analysis to evaluate the training's effectiveness and explore the influence of demographic variables. Ethical considerations, including informed consent and data confidentiality, will be strictly maintained.

This study is expected to provide valuable insights into the role of EI training in fostering resilience and mental health among Bangladeshi youth, contributing to healthier communities and informing future policy and program development.

ELIGIBILITY:
Inclusion Criteria:

1. being aged between 18 to 30 years
2. having a stable internet connection
3. agreeing to attend all four training sessions

Exclusion Criteria:

1. Previous experience in EI training
2. inability to attend the complete program
3. serious interruptions during the experiment

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 213 (Actual)
Dates: Start 2024-09-10 (Actual); Primary Completion 2024-10-10 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
Emotional Intelligence | 4 weeks
  Emotional Intelligence (EI) will be assessed via a self-report scale. The emotional intelligence scale was developed by Hyde, Pethe and Dhar in 2002. The Bengali version of the scale was subsequently adapted by Uzzaman and Karim in 2017. The scale typically consists of questions related to various aspects of emotional intelligence, with respondents indicating their level of agreement or frequency on a Likert scale. The total score (typically, ranging from 34-170) is used to determine overall emotional intelligence, with higher scores indicating greater EI. The original scale has a high degree of content validity. The scale has a split-half reliability of.88. The Bangla version of the Emotional Intelligence Scale had a Cronbach's alpha value of 0.92. With a mean of 0.58, all the item-total correlations were significant and ranged from 0.33-0.84. Convergent validity was also guaranteed by the Bangla version.

CONTACTS AND LOCATIONS:
Locations (1):
- Bangladesh Institute of Innovative Health Research, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: No
We do not plan to share Individual Participant Data (IPD) with other researchers. This decision is based on considerations such as participant privacy and confidentiality, the lack of explicit consent from participants for data sharing, and compliance with institutional or ethical guidelines. Protecting sensitive information remains our priority, and we aim to uphold the trust placed in us by our participants.

REFERENCES:
- [Background] Kotsou I, Nelis D, Gregoire J, Mikolajczak M. Emotional plasticity: conditions and effects of improving emotional competence in adulthood. J Appl Psychol. 2011 Jul;96(4):827-39. doi: 10.1037/a0023047. PMID 21443316
- [Background] World Medical Association. World Medical Association Declaration of Helsinki: ethical principles for medical research involving human subjects. JAMA. 2013 Nov 27;310(20):2191-4. doi: 10.1001/jama.2013.281053. No abstract available. PMID 24141714
- [Background] Durham MRP, Smith R, Cloonan S, Hildebrand LL, Woods-Lubert R, Skalamera J, Berryhill SM, Weihs KL, Lane RD, Allen JJB, Dailey NS, Alkozei A, Vanuk JR, Killgore WDS. Development and validation of an online emotional intelligence training program. Front Psychol. 2023 Aug 17;14:1221817. doi: 10.3389/fpsyg.2023.1221817. eCollection 2023. PMID 37663347
- [Background] Fernandez-Berrocal P, Extremera N. Emotional intelligence: a theoretical and empirical review of its first 15 years of history. Psicothema. 2006;18 Suppl:7-12. PMID 17295952
- [Background] Sekhri P, Sandhu M, Sachdev V. Emerging Understanding of Emotional Intelligence of Teenagers. Int J Clin Pediatr Dent. 2017 Jul-Sep;10(3):289-292. doi: 10.5005/jp-journals-10005-1452. Epub 2017 Feb 27. PMID 29104391
- [Background] Huffman JC, Niazi SK, Rundell JR, Sharpe M, Katon WJ. Essential articles on collaborative care models for the treatment of psychiatric disorders in medical settings: a publication by the academy of psychosomatic medicine research and evidence-based practice committee. Psychosomatics. 2014 Mar-Apr;55(2):109-22. doi: 10.1016/j.psym.2013.09.002. Epub 2013 Dec 25. PMID 24370112
- [Background] Goleman D. Emotional intelligence. İstanbul: Varlık Publication; 2001.
- [Background] Goleman D. Emotional intelligence: Why it can matter more than IQ for character, health and lifelong achievement. New York, NY: Bantam books; 1995.
- [Background] Erkuş A. Dictionary of psychological terms. Ankara: Doruk Publishing House; 1994.
- [Background] Mayer JD, Salovey P. What is emotional intelligence? In: Salovey P, Brackett MA, Mayer JD, editors. Emotional intelligence: Key readings on the Mayer and Salovey model, Dude Publishing; 2004, p. 29-59.